CLINICAL TRIAL: NCT05237401
Title: Survival of Molars With Degree III Periodontal Furcation Involvement Following Non-surgical or Surgical Therapy: a Multicentre Single-masked Superiority Randomised Controlled Trial.
Brief Title: Non-surgical vs. Surgical Therapy for Periodontal Furcations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 222112021
Record Dates: First submitted 2022-01-13; First posted 2022-02-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-10

CONDITIONS: Furcation Defects; Periodontitis; Surgical Procedure, Unspecified
MeSH Terms: conditions — Furcation Defects; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Surgical Periodontal treatment (NSPT) (Active Comparator): Half of the study participants (controls) will be randomised to receive continued non-surgical periodontal treatment (NSPT). All treatment will be carried out by the same therapist in each centre, including oral hygiene.
  Interventions: Procedure: Non-Surgical Periodontal treatment (NSPT)
- Surgical Periodontal treatment/ Open Flap Debridement (OFD) (Experimental): The other half of the study participants (test) will be randomised to receive surgical periodontal treatment in the form of open flap debridement (OFD). The aim of the surgery will be to achieve thorough debridement of the furcation area and (if possible) improve accessibility for patient-performed hygiene in the furcation area.
  Some of the included maxillary molars may have additional FI on the same tooth (for example, grade III FI buccal to mesial and grade I, II or III distal). In this occurrence, the other furcation will be treated according to judgment by the treating clinician. We anticipate that, based on inclusion criteria, the majority of cases will have multiple grade III FI.
  Interventions: Procedure: Surgical Periodontal treatment/ Open Flap Debridement (OFD)

INTERVENTIONS:
Procedure: Non-Surgical Periodontal treatment (NSPT) — participants will receive local anaesthesia, then thorough debridement of the root surface will be completed to the depth of the periodontal pocket and of the furcation lesion, by using sonic scaler (KaVo Sonicflex, KaVo, Germany), piezo-electric/ultrasonic devices with specific thin and delicate tips (such as Cavitron, Dentsply Sirona, US) and/or curettes.
  Arms: Non-Surgical Periodontal treatment (NSPT)
Procedure: Surgical Periodontal treatment/ Open Flap Debridement (OFD) — Patients will receive local anaesthesia and intrasulcular incisions will be made on the buccal and lingual/palatal aspects in order to reflect full-thickness flaps. After reflection of the flaps, the granulation tissue around the tooth will be removed with the non-cutting edge of a suitable scaling instrument such as a curette, taking care not to damage the root surfaces. Thorough debridement of the furcation area will be carried out by using diamond coated inserts, sonic scaler (KaVo Sonicflex, KaVo, Germany), piezo-electric/ultrasonic devices with specific thin and delicate tips (such as Cavitron, Dentsply Sirona, US) and/or curettes. Osteoplasty (removal of non-supporting bone) may be carried out, as judged by the operator. The surgical site will be closed with resorbable or non-resorbable sutures.
  Arms: Surgical Periodontal treatment/ Open Flap Debridement (OFD)

SUMMARY:
Periodontitis is an inflammatory disease of the tooth-supporting apparatus, which leads to attachment and bone loss and eventually to tooth loss if treatment is not provided.

When the periodontitis-related bone loss affects the area of root separation in molars, a furcation involvement (FI) is created. This represents a challenge in the treatment of periodontally-compromised molars, affecting the majority of patients with periodontitis. Based on a prevalence of severe forms of periodontitis in the UK and worldwide of about 10% of the population and on previous studies, we can assume that at least 5-10% of the general population are affected by FI.

Different treatment modalities are advocated for the treatment of FI, including non-surgical maintenance, resective (bone recontouring) and regenerative (reconstruction of bone and attachment) surgical treatments or tooth extraction. It has clearly emerged that FI at least doubles the risk of tooth loss. However, in the case of advanced through-and-through loss of attachment and bone in the furcation area (FI degree III), the clinician is often faced with a very difficult treatment decision, without being able to draw on much evidence from the literature. Interestingly, there are no randomised controlled trials exploring the most appropriate treatment for advanced furcation involvement. This has been highlighted in a recent systematic review commissioned by the European Federation of Periodontology.

DETAILED DESCRIPTION:
Subject recruitment All patients will be recruited from Periodontal Clinics at the participating centres in United Kingdom (Ravenscourt Dental Practice, 5 Ravenscourt avenue, Germany (University Hospital of Berlin, Bonn, Frankfurt and Greifswald), Sweden (Malmo), Spain (Santiago de Compostela), Italy (Torino) and Australia (Brisbane). When a potentially suitable patient is identified in the clinics, the assigned hospital consultant (or equivalent outside the UK) will inform him/her of the study and ask if the patient is interested in discussing this with a member of the research team. Then a member of the research team will approach the patient, provide more information about the study procedures and will give them an information sheet about the study. If the patient agrees to take part, they will be offered a baseline appointment. If they need more time to consider participation, they will be contacted by phone by a member of the periodontology research team within 1 week to enquire about their willingness to take part in the study and to give them the opportunity to ask any questions about the study. If all inclusion/exclusion criteria cannot be verified at the new patient clinic appointment, a review appointment prior to baseline will be offered. Each subject will be part of the study for approximately 5 years.

At the time of subject recruitment in addition to information about the study; the overall management plan will be discussed with the patient. The responsible consultant (or equivalent) will provide information about the treatment of the non-study sites and what additional treatment will be provided for those areas. This will commence once the study sites have been treated. If any other dental treatment is required before the baseline visit (e.g. fillings or extractions), as judged by the responsible consultant (or equivalent), such treatment will be carried out prior to baseline.

Screening Procedures Potential new patients which may be suitable for the study will be screened alongside all other patients attending Periodontology clinics at the participating centres and accepted based upon the inclusion and exclusion criteria above.

Randomisation Procedures Randomisation for test or control treatment will be carried out between baseline (visit 1) and visit 2. The randomisation service 'Sealed envelope' will be used in each centre for randomisation and to ensure allocation concealment. A sealed envelope will be enclosed with the patient's notes by personnel not directly involved in the study. The therapist will be informed about treatment allocation by opening the envelope at the beginning of the treatment appointment.

For each centre patients will be allocated to the two treatment groups using a randomisation list that was previously prepared by the study statistician. For important influencing factors ('centre') stratified randomisation will be carried out as recommended , especially in case of small sample sizes.

Clinical periodontal examination Dichotomous (no/yes) full mouth plaque scores (FMPS) will be recorded, identifying tooth surfaces revealing the visual presence of plaque following the use of plaque-disclosing tablets. Periodontal measurements will be taken by the calibrated examiner at six sites per tooth using a manual University of North Carolina (UNC-15) periodontal probe. The following periodontal measurements will be taken full mouth at 6 sites per tooth: probing pocket depth (PPD), recession of the gingival margin from the cemento-enamel junction (CEJ), dichotomous (no/yes) bleeding on probing (BoP) . Recession will be recorded as a negative number if the gingival margin is above CEJ (or the assigned reference e.g. restorative margin); and as a positive number (incl. 0) if margin is on (0) or below CEJ (>0). Further, tooth mobility (no/yes and degree 1, 2 or 3, horizontal furcation involvement using a Nabers probe (no/yes and degree 1, 2 or 3) and finally vertical furcation involvement (no/yes and class A, B or C) measured with a UNC-15 probe will be recorded. Clinical attachment levels (CAL) will be calculated as PPD + recession. The amount of keratinized gingiva by the test furcation will be recorded. This is part of standard care.

Sub-gingival plaque sampling

Sub-gingival plaque samples will be collected from:

* test site (TS): preferably buccal surface of furcation site; alternatively, mesial furcation site in maxillary furcation if buccal furcation is not degree III
* control site (CS): ideally, symmetrical contralateral site in case of no furcation involvement. Alternatively, another site with PPD<4mm and no bleeding on probing will be chosen and recorded.

For example, LR6 buccal (furcation III) as test site and LL6 buccal (no FI) as control site. Plaque samples will be collected from the selected TS and CS at baseline and then following treatment at 4 months, at 8 months, at 12 months and at all subsequent 12-monthly follow-ups (a total of 8 time-points).

Ahead of the sampling procedure, the supra-gingival plaque will be carefully removed, the site isolated with cotton rolls and gently dried. A sterile curette will then be inserted to the bottom of the pocket and removed after a single stroke and the content will be placed in a test tube containing a buffer solution such as TE buffer solution (Cat No. 93283 Sigma-Aldrich) and stored at -80ºC until the time of analysis. The aim of taking sub-gingival plaque samples at these time points is to assess the composition of the sub-gingival microbiota before and after treatment in test and control sites.

Data Recording/Reporting The results of the laboratory analyses will be recorded in encrypted databases according to standard procedures.

Adverse Events (AE) An AE is any untoward medical occurrence in a subject to whom a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporarily associated with study activities.

Notification and reporting Adverse Events or Reactions If the AE is not defined as SERIOUS, the AE is recorded in the study file and the participant is followed up by the research team. The AE is documented in the participants' medical notes (where appropriate) and the CRF.

Statistical analyses Comprehensive descriptive analyses will be done for primary and secondary endpoints. Time trajectories of primary and secondary endpoints within treatment groups will be graphically assessed. Also, distributions of primary and secondary endpoints within groups over time points will be graphically shown.

The analysis level is the tooth (one target molar per patient is included). In case of more than 1 suitable molar per patient, the 'study molar' will be chosen based on deepest PPD (or deepest CAL in case of same PPD).

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 teeth present
* Diagnosis of Severe Periodontitis stage III or IV
* At least one maxillary/ mandibular molar with: i) degree III horizontal furcation involvement (at least between 2 roots for maxillary molars) , ii) class B vertical furcation involvement (bone loss up to the middle third of root cones), iii) residual probing pocket depths > 5 mm in furcation area, iv) maximum mobility degree Iand v) not already accessible for self-performed oral hygiene
* Received a course of non-surgical periodontal therapy within the past six months

Exclusion Criteria:

Patient:

* Full mouth plaque score > 30%
* A course of antibiotics within the past 3 months
* Pregnant/lactating women
* Relevant medical history as evaluated by the examining clinician which may have the potential to affect periodontal surgical treatment
* Individuals on long-standing (2 or above years) supportive periodontal therapy (SPT) management plans

Molar affected by FI:

* Ongoing endodontic pathology affecting the furcation involved molar, as judged by the examining clinician
* Previous periodontal surgical treatment to the furcation affected molar within the previous 5 years
* Endodontically treated molar tooth without a full coverage restoration
* 'Unrestorable' molar tooth (lacking adequate tooth structure to provide a restoration) as deemed by the examining clinician.
* Molar tooth acting as a bridge abutment
* The presence of occlusal dysfunction as assessed by the examining clinician

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
5-year tooth survival | 5 years
  to test the survival of the tooth with advanced furcation after 5 years

SECONDARY OUTCOMES:
Maximum Pocket depth (PPD) | 5 years
  in mm at 5 years (tooth level; maximum over 6 sites per tooth)
Maximum Clinical attachment level CAL | 5 years
  in mm at 5 years (tooth level; maximum over 6 sites per tooth)
Radiographic bone levels | 5 years
  tooth level, measured radiographically
Patient's discomfort measurement | 5 years
  measured with patient questionnaires at 5 years
Time needed for each study appointment during maintenance therapy | 5 years
  to evaluate the efficiency of routine dental hygiene
Cost-effectiveness Analysis | 5 years
  The costs will be collected from the perspective of the health insurance party payer.The effectiveness measure will be the tooth retention time (years in function)
Cost-Utility analyses | 5 years
  The costs will be collected from the perspective of the health insurance party payer. A questionnaire (OHIP-14) will be used as utility value in additional cost ultility analyses.
Occurrence of root caries in furcation area | 5 years
  yes/no answer for presence or absence of caries
1-year tooth survival | 1 year
  to test the survival of the tooth with advanced furcation after 12 months
3-year tooth survival | 3 years
  to test the survival of the tooth with advanced furcation after 36 months
Microbiological analysis | 1 year
  Plaque microbiome will be quantitative and qualitative analysed using the shot-gun metagenomic analysis based on DNA extraction and subsequent analysis.
Microbiological analysis | 5 years
  Plaque microbiome will be quantitative and qualitative analysed using the shot-gun metagenomic analysis based on DNA extraction and subsequent analysis.
Fractures | 5 years
  yes/no index to assess root fracture long term
Endodontic complications | 5 years
  accessory canals in the furcation or mid-root region as a route for bacterial infection the pulp tissue
Tooth mobility | 5 years
  to assess the grade of tooth mobility with a (yes/no) index
Further treatment needed | 5 years
  yes/no index assessing the need for repeated instrumentation and/or prosthetic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, Study Chair — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No